CLINICAL TRIAL: NCT00381472
Title: A Phase III, Randomised, Double-blind, Placebo-controlled, Parallel Group Study of Six Months Treatment With Ropinirole CR as Adjunctive Therapy in Patients With Parkinson's Disease Who Are Not Optimally Controlled on L-dopa
Brief Title: Investigational Parkinson's Disease In Patients Not Well Controlled On L-dopa
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 101468/169
Record Dates: First submitted 2006-09-26; First posted 2006-09-27 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Dyskinesia; Adjunctive Therapy with L-dopa
MeSH Terms: conditions — Parkinson Disease; Dyskinesias | interventions — ropinirole

INTERVENTIONS:
Drug: Ropinirole

SUMMARY:
The purpose of this double-blind, placebo controlled study is to evaluate the safety and effectiveness of an investigational Parkinson's disease drug in patients with advanced disease who are not well-controlled on their L-dopa medication.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease
* Modified Hoehn and Yahr Scale Stages II - IV
* Stable dose of L-dopa for at least 4 weeks prior to screening.
* Lack of control with L-dopa therapy.
* Women of child-bearing potential must use a clinically accepted form of birth control.

Exclusion Criteria:

* Significant and/or uncontrolled medical conditions (excluding Parkinson's disease) within 3 months of screening.
* Any abnormality, at screening, that is considered clinically relevant by the Investigator.
* Dementia
* Use of dopamine agonists within 4 weeks of screening visit.
* Participation in other investigational drug studies.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 393
Dates: Start 2003-06; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Mean change from baseline in awake time "off" at Week 24 LOCF (last observation carried forward).

SECONDARY OUTCOMES:
Mean change from baseline in:
amount and percent of awake time spent "on"
percent awake time spent "off"
Unified Parkinson's Disease Rating Scale (UPDRS) total motor score
UPDRS Activities of Daily Living score

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (64):
- United States (27):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Northridge, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Englewood, Colorado
  - GSK Investigational Site, Boca Raton, Florida
  - GSK Investigational Site, Panama City, Florida
  - GSK Investigational Site, St. Petersburg, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Atlanta, Georgia
  - GSK Investigational Site, Augusta, Georgia
  - GSK Investigational Site, Glenview, Illinois
  - GSK Investigational Site, Kansas City, Kansas
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Bingham Farms, Michigan
  - GSK Investigational Site, Southfield, Michigan
  - GSK Investigational Site, Traverse City, Michigan
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Albany, New York
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Toledo, Ohio
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Upland, Pennsylvania
  - GSK Investigational Site, Wichita Falls, Texas
  - GSK Investigational Site, Milwaukee, Wisconsin
- Belgium (5):
  - GSK Investigational Site, Antwerp
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Hasselt
  - GSK Investigational Site, Leuven
  - GSK Investigational Site, Roeselare
- Czechia (6):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
- France (4):
  - GSK Investigational Site, Aix-en-Provence
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Poitiers
- Germany (2):
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony
- Hungary (4):
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Vasvari Pal Street 2, H=9023 Gyor
- Italy (5):
  - GSK Investigational Site, Pozzilli (IS), Molise
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Grosseto, Tuscany
  - GSK Investigational Site, Lido Di Camaiore (LU), Tuscany
  - GSK Investigational Site, Vicenza, Veneto
- Poland (10):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Cibórz
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Leszno
  - GSK Investigational Site, Lublin
  - GSK Investigational Site, Szwajcarska 3
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
- GSK Investigational Site, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] B P Hersh, S A Factor, L Giorgi Ropinirole 24-hour prolonged release improves motor function and activities of daily living as an adjunct to L-dopa in Parkinson's Disease. Eur J Neurol. September 2006/Suppl 2: 13/S2-P2202
- [Background] F Stocchi, B Hersh, N Earl, B Scott Safety and tolerability of ropinirole 24-hour prolonged release in patients with early and advanced Parkinson's Disease. Movement Disorders, November 2006; 21 (Suppl.15) S572/P894.
- [Background] F Stocchi, M A Stacy, L Giorgi, N L Earl Safety and tolerability of ropinirole 24-hour prolonged release as adjuctive therapy to L-dopa in patients with Parkinson's Disease. Eur J Neurol. September 2006/Suppl 2-13/a2P2201
- [Background] Reichmann H, Cooper J, Rolfe K, Martinez-Martin P. Sleep Duration and "on" Time during Different Periods of the Day and Night in Patients with Advanced Parkinson's Disease Receiving Adjunctive Ropinirole Prolonged Release. Parkinsons Dis. 2011;2011:354760. doi: 10.4061/2011/354760. Epub 2011 May 11. PMID 21687750
- [Background] Ray Chaudhuri K, Martinez-Martin P, Rolfe KA, Cooper J, Rockett CB, Giorgi L, Ondo WG. Improvements in nocturnal symptoms with ropinirole prolonged release in patients with advanced Parkinson's disease. Eur J Neurol. 2012 Jan;19(1):105-13. doi: 10.1111/j.1468-1331.2011.03442.x. Epub 2011 Jun 23. PMID 21699627
- [Background] K Sethi, N Earl, R Hauser Ropinirole 24-hour prolonged release improves disease-specific and global symptoms when used as adjunctive therapy to L-dopa in patients with advanced Parkinson's Disease. Movement Disorders, November 2006; 21 (Suppl.15) S570/P887
- [Background] M A Stacy, K D Sethi, N L Earl Ropinirole 24-hour prolonged release improves sleep but does not increase daytime sleepiness when used as adjunctive therapy in patients with Parkinson's Disease not optimally controlled by L-dopa. Movement Disorders, November 2006 S15/9.21:1543-1559
- [Background] M Stacy, R Pahwa, N Earl Ropinirole 24-hour prolonged release reduces "off" time and reduces the need for L-dopa when used as adjunctive therapy in patients with advanced Parkinson's Disease Movement Disorders, November 2006: 21 (Suppl 15) S596/P972
- [Background] R A Hauser, M A Stacy, B P Hersh Ropinirole 24 hour prolonged release reduces off time and improves depression when used as adjunctive therapy in patients with Parkinson's disease not optimally controlled with L-dopa Movement Disorders S15-21-P8
- [Background] R Pahwa, F Stocchi, M A Stacy Ropinirole 24-hour prolonged release is effective in sparing L-dopa dose and improving symptoms as adjuctive therapy in Parkinson's Disease. Eur J Neurol, September 2005/Suppl 2:s2-P2203
- [Background] R Pahwa, M Stacy, E Elmer, S Isaacson Ropinirole 24-hour prolonged release provides efficacy as early as Week 2 when used as adjunctive therapy to L-dopa in patients with advanced Parkinson's Disease Movement Disorders, November 2006: 21 (Suppl 15) S595/P968.
- [Background] Pahwa R, Stacy MA, Factor SA, Lyons KE, Stocchi F, Hersh BP, Elmer LW, Truong DD, Earl NL; EASE-PD Adjunct Study Investigators. Ropinirole 24-hour prolonged release: randomized, controlled study in advanced Parkinson disease. Neurology. 2007 Apr 3;68(14):1108-15. doi: 10.1212/01.wnl.0000258660.74391.c1. PMID 17404192
- [Background] R Pahwa, S Factor, L Elmer Ropinirole 24 hour prolonged release reduces awake time spent "off" in patients with Parkinson's disease not optimally controlled with L-dopa. Neurology, April 2006. 66 (Suppl 2): A292. P05.135
- [Background] R Pahwa, SA Factor, L Elmer Ropinirole 24 hour prolonged release reduces "off" time in patients with Parkinson's disease not optimally controlled with L-dopa. Eur J Neurol, September 2006/Suppl2, 13/s2:P2154.
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 101468/169 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register